CLINICAL TRIAL: NCT04501237
Title: Efficacy of Sleep Hygiene Measures in the Occurrence of Sleep Bruxism in Children
Brief Title: Sleep Hygiene Measures for Sleep Bruxism in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of Pelotas (Other)
Responsible Party: Principal Investigator, Maximiliano Sergio Cenci, Professor, Federal University of Pelotas
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PPGO 032
Record Dates: First submitted 2020-08-03; First posted 2020-08-06 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2020-08

CONDITIONS: Sleep Bruxism, Childhood
MeSH Terms: conditions — Sleep Bruxism

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bruxers without sleep hygiene instructions (No Intervention)
- Bruxers with sleep hygiene instructions (Experimental)
  Interventions: Behavioral: Bruxers with sleep hygiene instructions

INTERVENTIONS:
Behavioral: Bruxers with sleep hygiene instructions — the test group will receive instructions of sleep hygiene, limited use of screens and a relaxation audio.
  Arms: Bruxers with sleep hygiene instructions

SUMMARY:
The aim of the study is to evaluate the efficacy of sleep hygiene measures for the possible improvement of sleep bruxism in children through a randomized controlled clinical study of children under 8 years of age with probable sleep bruxism. In randomization both groups will receive information about bruxism, and the test group will receive instructions of sleep hygiene, limited use of screens and a relaxation audio. The occurrence of sleep bruxism will be assessed through a diary to be completed by the child's responsible party. A randomized, stratified sample of approximately 16 children will be included in the study. One group will be composed of 8 children with probable sleep bruxism who will receive the sleep hygiene intervention, and another group of children who will only receive instructions on sleep bruxism, with causes and consequences. Participants will be followed-up for 30 days. Parents will respond to a questionnaire about socioeconomic, demographic (child's age and gender), as well as parafunctional habits such as nail biting, biting objects, pacifier sucking, finger / thumb sucking and bottle feeding, child's sleep characteristics, screen habits, parental smoking, problems breathing, parental profession and also on psychological issues. Sleep habits will also be answered in this questionnaire, and parents will also answer the Strengths and Difficulties Questionnaire. The children over 6 years old will respond a Child Stress Scale and the Child of stressing sources in child; children less than 6 years will have the questionnaire responded by parents. The children will undergo a clinical examination to assess dental wear, according to the BEWE (Basic Erosive Wear Examination Index). The study evaluations consist of baseline, 1, 7, 15 and 30 days.

ELIGIBILITY:
Inclusion Criteria:

* children with probable sleep bruxism

Exclusion Criteria:

* systemic diseases;
* Medical and/or behavioral conditions that requires special considerations regarding management/treatment of the child.

Ages: 2 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2021-02-01 (Estimated); Study Completion 2021-05-01 (Estimated)

PRIMARY OUTCOMES:
Questionnaire | Responded 1 month after intervention in both groups
  Strengths and Difficulties Questionnaire

SECONDARY OUTCOMES:
Clinical evaluation of child teeth | Analyzed 1 month after intervention in both groups
  Basic Erosive Wear Examination Index

CONTACTS AND LOCATIONS:
Locations (1):
- School of dentistry, Pelotas, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided